CLINICAL TRIAL: NCT00280592
Title: Prospective, Randomized, Double-blind, Placebo-controlled Study on Parallel Groups Evaluating the Efficacy and Safety of Cranberry (Vaccinium Macrocarpon) in Prevention of Urinary Tract Infections in Multiple Sclerosis Patients.
Brief Title: Cranberry for Prevention of Urinary Tract Infections in Multiple Sclerosis Patients
Acronym: CANNEBERGE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Collaborators: Pierre Fabre Laboratories (Industry); Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: AFSSAPS 051016; PHRC/04-03 (Other: Rennes University Hospital); CIC0203/039
Record Dates: First submitted 2006-01-20; First posted 2006-01-23 (Estimated); Last update posted 2012-05-21 (Estimated); Status verified 2008-05

CONDITIONS: Multiple Sclerosis; Urinary Tract Infections; Bladder Dysfunction
Keywords: Prophylaxis; Cranberry; Neurogenic bladder
MeSH Terms: conditions — Multiple Sclerosis; Urinary Tract Infections; Urinary Bladder, Neurogenic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Cranberry (Experimental): Cranberry
  Interventions: Drug: Cranberry

INTERVENTIONS:
Drug: Cranberry — Dry essence of cranberry presented as 18 mg of proanthocyanidines sachets of powdered cranberry. Cranberry juice is administered twice a day (in the morning and in the evening).
  Other Names: Vaccinium macrocarpon
  Arms: Cranberry
Drug: Placebo — Placebo presented as sachets of powder. Placebo juice is administered twice a day (in the morning and in the evening).
  Arms: Placebo

SUMMARY:
Bladder dysfunction occurs at some time in most patients with multiple sclerosis and these patients are prone to have recurrent urinary tract infections. Cranberry has been traditionally used for the treatment and prophylaxis of urinary tract infections but there is no reliable randomized controlled trial demonstrating evidence of cranberry's utility in this disease. The aim of our study is to assess the efficacy and safety of cranberry in the prophylaxis of urinary tract infections in patients with multiple sclerosis with a prospective randomized, double-blind and placebo-controlled clinical trial.

DETAILED DESCRIPTION:
Bladder dysfunction occurs at some time in 70 to 90% of patients with multiple sclerosis and these patients are prone to have recurrent urinary tract infections (UTI), leading to an important morbidity. Cranberry has been traditionally used for the treatment and prevention of UTI and research suggests that its mechanism of action is preventing bacterial adherence to host cell surface membrane.

However, systematic reviews show the small sample sizes and the poor quality of available trials, determining that there is no reliable evidence of effectiveness of cranberry in UTI prophylaxis. Therefore, to assess whether cranberry is effective in reducing UTI in patients with multiple sclerosis, we have designed a randomized, double-blind, placebo-controlled trial. Efficacy will be evaluated on the time to onset of a UTI in the first year of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 70, with multiple sclerosis, neurologically stable for at least 3 months
* With an EDSS score ≥ 3
* Symptomatic bladder dysfunction: frequency, urgency, dysuria, incontinence (at least one of these symptoms), needing intermittent catheterization or not
* Ambulatory at inclusion
* Able to undergo evaluation
* Informed written consent

Non-inclusion Criteria:

* Regular consumption of cranberry within 3 months before inclusion
* Symptomatic urinary tract infection at inclusion
* Chronic renal failure (creatinin clearance < 10ml/min)
* Patients with urinary permanent catheterization
* Patients with hyperuricemia and risk of uric acid lithiasis
* Patients with oral anticoagulant treatment (antivitamins K)
* Peptic ulcer
* Intolerance to cranberry and/or excipients
* Urinary tract infections antibioprophylaxis

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 2006-01; Primary Completion 2008-03 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Time to onset of a first UTI within one year of treatment. | one year

SECONDARY OUTCOMES:
Rate of patients with at least one UTI during the one-year treatment | Determined at M3, M6, M9 and M12
Number of UTI | Determined at M3, M6, M9 and M12
Score on Qualiveen® scale | Determined at M3, M6, M9 and M12
Symptomatology of urinary disorders | Determined at M3, M6, M9 and M12
EDSS score | Determined at M3, M6, M9 and M12
Number of multiple sclerosis attacks | Determined at M3, M6, M9 and M12
Antibiotics consumption | Determined at M3, M6, M9 and M12
Safety of cranberry | Determined at M3, M6, M9 and M12
Patients' observance to treatment | Determined at M3, M6, M9 and M12

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Michel Reymann, PhD, Study Chair — CHU Rennes; Philippe Gallien, MD, Principal Investigator — CHU Rennes
Locations (10):
- France (10):
  - Unité de Médecine Physique et Réadaptation - CHU Jean Minjoz, Besançon
  - Service de Médecine Physique et Réadaptation - Hôpital Pellegrin, Bordeaux
  - Service de Médecine Physique et Réadaptation - Hôpital Raymond Poincaré, Garches
  - Consultations maladies infectieuses et tropicales, Hôpital Raymond Poincaré, Garches
  - Médecine Physique et Réadaptation - Groupe Hospitalier de l'institut Catholique de Lille - Hôpital Saint Philibert, Lomme
  - Rééducation Neurologique et Explorations Périnéales - Hôpital Rothschild, Paris
  - Centre Mutualiste de Rééducation et de Réadaptation Fonctionnelles de KERPAPE, Ploemeur
  - Service de Médecine Physique et Réadaptation - Hôpital Pontchaillou, Rennes
  - Centre de Médecine Physique et Réadaptation Notre Dame de Lourdes, Rennes
  - Service de médecine physique et réadapation Hopital de Rangueil, Toulouse

REFERENCES:
- [Derived] Williams G, Stothart CI, Hahn D, Stephens JH, Craig JC, Hodson EM. Cranberries for preventing urinary tract infections. Cochrane Database Syst Rev. 2023 Nov 10;11(11):CD001321. doi: 10.1002/14651858.CD001321.pub7. PMID 37947276
- [Derived] Williams G, Hahn D, Stephens JH, Craig JC, Hodson EM. Cranberries for preventing urinary tract infections. Cochrane Database Syst Rev. 2023 Apr 17;4(4):CD001321. doi: 10.1002/14651858.CD001321.pub6. PMID 37068952
- [Derived] Gallien P, Amarenco G, Benoit N, Bonniaud V, Donze C, Kerdraon J, de Seze M, Denys P, Renault A, Naudet F, Reymann JM. Cranberry versus placebo in the prevention of urinary infections in multiple sclerosis: a multicenter, randomized, placebo-controlled, double-blind trial. Mult Scler. 2014 Aug;20(9):1252-9. doi: 10.1177/1352458513517592. Epub 2014 Jan 8. PMID 24402038